CLINICAL TRIAL: NCT01986114
Title: A Long-Term Study of SM-13496 in Patients With Bipolar I Disorder.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1002002; JapicCTI-132319 (Registry Identifier: JAPIC Clinical Trials Information); 2013-003039-31 (EudraCT Number)
Record Dates: First submitted 2013-11-04; First posted 2013-11-18 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Bipolar I Disorder
MeSH Terms: interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SM-13496 20-120mg (Experimental): once daily orally SM-13496 20-120 mg flexibly dosed
  Interventions: Drug: SM-13496

INTERVENTIONS:
Drug: SM-13496
  Other Names: Lurasidone

SUMMARY:
The study evaluates the long-term efficacy and safety of SM-13496 in patients with bipolar I disorder.

DETAILED DESCRIPTION:
The study objective is to evaluate the long-term efficacy and safety of SM-13496 (20-120 mg/day) in patients with bipolar I disorder.

ELIGIBILITY:
Inclusion Criteria:

Patients who completed the D1002001 study

・Patients who completed the D1002001 study and who are considered by the investigator to be eligible and without safety concerns.

Patients who did not participate in the D1002001 study

* Patients who were fully informed of and understand the objectives, procedures, and possible benefits and risks of the study and who provided written voluntary consent to participate in the study.
* Outpatients aged 18 through 74 years at the time of consent
* Patients meets DSM-IV-TR criteria for bipolar I disorder, most recent episode manic, hypomanic, or mixed with or without rapid cycling disease course (≥ 4 episodes of mood disturbance, but < 8 episodes in the previous 12 months prior to screening).

Exclusion Criteria:

* Patients with imminent risk of suicide or injury to self, others, or property.
* Patients who are otherwise considered ineligible for the study by the investigator.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2014-01-29 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2018-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director, Drug Development Division, Study Director — Sumitomo Pharma Co., Ltd.
Locations (8):
- Japan 68 sites, Tokyo, Japan
- Lithuania 3 sites, Kaunas, Lithuania
- Malaysia 5 sites, Kuala Lumpur, Malaysia
- Philippines 5 sites, Manila, Philippines
- Russia 19 sites, Moscow, Russia
- Slovakia 5 sites, Žilina, Slovakia
- Taiwan 8 sites, Taipei, Taiwan
- Ukraine 9 sites, Kiev, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Higuchi T, Kato T, Miyajima M, Watabe K, Masuda T, Hagi K, Ishigooka J. Lurasidone in the long-term treatment of Japanese patients with bipolar I disorder: a 52 week open label study. Int J Bipolar Disord. 2021 Aug 2;9(1):25. doi: 10.1186/s40345-021-00230-8. PMID 34342746
- [Derived] Ishigooka J, Kato T, Miyajima M, Watabe K, Masuda T, Hagi K, Higuchi T. Lurasidone in the Long-Term Treatment of Bipolar I Depression: A 28-week Open Label Extension Study. J Affect Disord. 2021 Feb 15;281:160-167. doi: 10.1016/j.jad.2020.12.005. Epub 2020 Dec 8. PMID 33321381

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 495 represents the total number of subjects who were treated with study drug.
Groups:
- SM-13496 20-120mg: once daily orally
  SM-13496 (lurasidone HCl): SM-13496 20-120mg
Period: Overall Study
Arm/Group | SM-13496 20-120mg
Started | 495
Completed | 339
Not Completed | 156
Not completed — Adverse Event | 59
Not completed — Lack of Efficacy | 23
Not completed — Withdrawal by Subject | 58
Not completed — Noncompliance | 3
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 5
Not completed — Other reason | 7

BASELINE CHARACTERISTICS:
Population: Safety population-received at least one dose of study medication
Arm/Group | SM-13496 20-120mg
Number analyzed (Participants) | 495
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (12.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 259
  Male | 236
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 225
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 270
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Japan | 199
  Philippines | 8
  Taiwan | 7
  Ukraine | 117
  Malaysia | 11
  Slovakia | 15
  Lithuania | 9
  Russia | 129

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With at Least One Adverse Event (AE) and Adverse Drug Reaction (ADR)
Description: The number and percentage of subjects with at least one adverse event and adverse drug reaction
Time Frame: 28, 52 weeks
Measure: Count of Participants; unit: Participants
Groups:
- SM-13496 20-120mg (Overall, 28 Weeks): once daily orally
  SM-13496 (lurasidone HCl): SM-13496 20-120mg flexibly dosed up to 28 weeks
- SM-13496 20-120mg (Japan, 52 Weeks): once daily orally
  SM-13496 (lurasidone HCl): SM-13496 20-120mg flexibly dosed up to 52 weeks
Arm/Group | SM-13496 20-120mg (Overall, 28 Weeks) | SM-13496 20-120mg (Japan, 52 Weeks)
Number analyzed (Participants) | 495 | 199
Participants | 352 | 169

2. Secondary Outcome: Change From Long Term Study Baseline to LOCF Endpoint in the Montgomery-Asberg Depression Rating Scale (MADRS) Score
Description: Montgomery-Asberg Depression Rating Scale (MADRS)is a clinician-rated assessment of a subject's level of depression.
  The MADRS total score ranges from a minimum of 0 to a maximum of 60. For the MADRS total score, low scores indicate a better outcome and high scores indicate a worse outcome. When change from baseline is considered, a negative (decrease in score) value is considered a better outcome, and a positive (increase in score) value is considered a worse outcome.
  The MADRS contains ten (10) items. The total score is computed as the sum of the scores for the 10 items.
Time Frame: Baseline, 52 weeks and each month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SM-13496 20-120mg (Overall, 28 Weeks) | SM-13496 20-120mg (Japan, 52 Weeks)
Number analyzed (Participants) | 494 | 198
units on a scale | -4.4 (12.09) | 1.1 (12.58)

3. Secondary Outcome: Change From Long Term Study Baseline to LOCF Endpoint in the Young Mania Rating Scale (YMRS) Total Score.
Description: YMRS (Young Mania Rating Scale) is a clinician-rated assessment of the severity of mania in subjects with a diagnosis of bipolar disorder.
  The YMRS total score ranges from a minimum of 0 to a maximum of 60. For the YMRS total score, low scores indicate a better outcome and high scores indicate a worse outcome. When change from baseline is considered, a negative (decrease in score) value is considered a better outcome, and a positive (increase in score) value is considered a worse outcome.
  The YMRS contains eleven (11) items. The total score is computed as the sum of the scores for the 11 items.
Time Frame: Baseline, 52 weeks and each month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SM-13496 20-120mg (Overall, 28 Weeks) | SM-13496 20-120mg (Japan, 52 Weeks)
Number analyzed (Participants) | 494 | 198
units on a scale | -1.0 (4.54) | -2.0 (6.73)

4. Secondary Outcome: Number of Subjects Who Experienced Recurrence/Relapse of Any Mood Event From Clinical Stability of Bipolar Disorder.
Description: The number and percentage of subjects who experienced recurrence/relapse of any mood event from clinical stability of bipolar disorder.
Time Frame: Baseline to 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | SM-13496 20-120mg (Overall, 28 Weeks) | SM-13496 20-120mg (Japan, 52 Weeks)
Number analyzed (Participants) | 495 | 199
Participants | 14 | 18

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 28 weeks (outside Japan) and 52 weeks (Japan).
Arm/Group | SM-13496 20-120mg (Overall, 28 Weeks) | SM-13496 20-120mg (Japan, 52 Weeks)
All-Cause Mortality (participants affected / at risk) | 0/495 | 0/199
Serious Adverse Events (participants affected / at risk) | 19/495 | 12/199
Other Adverse Events (participants affected / at risk) | 250/495 | 137/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SM-13496 20-120mg (Overall, 28 Weeks) (N=495) | SM-13496 20-120mg (Japan, 52 Weeks) (N=199)
Disease progression (General disorders) | 8 (8) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1) | 1 (1)
Glucose urine present (Investigations) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Akathisia (Nervous system disorders) | 1 (1) | 1 (1)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1) | 1 (1)
Alcoholism (Psychiatric disorders) | 1 (1) | 1 (1)
Hallucination, auditory (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 1 (1) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 3 (3) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SM-13496 20-120mg (Overall, 28 Weeks) (N=495) | SM-13496 20-120mg (Japan, 52 Weeks) (N=199)
Diarrhoea (Gastrointestinal disorders) | 14 (15) | 10 (11)
Nausea (Gastrointestinal disorders) | 35 (38) | 24 (25)
Vomiting (Gastrointestinal disorders) | 17 (21) | 13 (13)
Disease progression (General disorders) | 16 (17) | 10 (11)
Nasopharyngitis (Infections and infestations) | 51 (63) | 53 (72)
Weight increased (Investigations) | 31 (31) | 17 (17)
Akathisia (Nervous system disorders) | 91 (104) | 60 (64)
Dystonia (Nervous system disorders) | 13 (15) | 10 (11)
Headache (Nervous system disorders) | 37 (46) | 16 (19)
Parkinsonism (Nervous system disorders) | 34 (43) | 15 (25)
Somnolence (Nervous system disorders) | 41 (44) | 24 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-03-15): https://cdn.clinicaltrials.gov/large-docs/14/NCT01986114/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT01986114/SAP_001.pdf